CLINICAL TRIAL: NCT00315289
Title: A Prospective Study of Primary Surgical Treatment of Nasolacrimal Duct Obstruction in Children Less Than Four Years Old
Brief Title: Study of Primary Surgical Treatment of Nasolacrimal Duct Obstruction in Children Less Than Four Years Old
Acronym: NLD1
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Jaeb Center for Health Research
Other Study IDs: NEI-116; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-01

CONDITIONS: Nasolacrimal Duct Obstruction
Keywords: Nasolacrimal duct obstruction; Simple probing; Balloon catheter dilation; Nasolacrimal intubation
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Nasolacrimal balloon catheter duct dilation
Procedure: Nasolacrimal intubation
Procedure: Simple Nasolacrimal duct probing

SUMMARY:
The purpose of this study is:

* To report the success proportions of simple probing within different age groups of patients under 24 months of age.
* To obtain descriptive data regarding symptoms and quality of life in patients receiving simple probing.
* To obtain similar data for simple probing in patients 24 months of age or older, for intubation in patients age 6 - <48 months, and for balloon catheter dilation in patients age 6 - <48 months.

DETAILED DESCRIPTION:
Nasolacrimal duct obstruction (NLDO) is a common ocular condition in the first year of life. Most cases will resolve spontaneously or with massage. Many studies of primary treatment of nasolacrimal duct obstruction have been reported. These case series have largely been retrospective, uncontrolled, and conducted in single centers.

Simple probing is the most widely-used initial treatment for NLDO in infancy. Two differing approaches to simple probing have been most often been used, immediate office probing (early probing-generally after 6 months of age), and medical management (episodic antibiotic drops with massage of the lacrimal sac) until 9-13 months of age followed by probing under general anesthesia (late probing). The possible advantages of early probing are the avoidance of general anesthesia, immediate resolution of symptoms, lesser cost, and prevention of fibrosis from inflammation in the nasolacrimal duct. The advantages of late probing include more comfort with the procedure and the avoidance of the procedure completely. Both early and late probing approaches are usually successful for treatment of NLDO in patients under 2 years of age, with reported success proportions varying from between 54% to 98%. Although a number of studies have found that probing was highly successful and without an age-related decline until at least 4 years of age and beyond, there is a suspicion among other clinicians of a clinically-important decline in the success proportions among progressively older age groups of preschool children. A large prospective interventional case series might help to clarify whether there is an age-related decline in success.

Balloon catheter dilation has become popular for the initial surgical treatment of NLDO especially in children older than one year. This procedure involves probing of the nasolacrimal duct with a semiflexible wire probe with an inflatable balloon on the tip.

Nasolacrimal intubation has been used for primary treatment by clinicians in older children or when the duct feels tight. While generally successful, there is less certainty of the success proportions for this procedure when performed as a primary treatment. It is also unknown how often this procedure is used for initial treatment.

Probing of the nasolacrimal duct for the repair of NLDO is a very successful procedure in infancy and childhood. Simple probing has long been the standard approach, though the age at which the procedure declines in effectiveness is controversial. Clinicians have been urged by manufacturers of medical equipment to consider intubation and balloon dilation even in the age range in which probing is highly successful, to further increase the chance of success.

A prospective non-randomized study of the outcomes from many centers of all strategies might allow better estimates of success for the techniques most often used over an extended age range. Such a study might help to define factors associated with failure of each of the techniques.

The study has been designed as an observational study that approximates standard clinical practice. All procedures are consistent with standard care with the exception of a questionnaire which the patient's parent will complete at each study visit on NLDO symptoms and quality of life. The surgical center is not engaged in the research and no data will be collected by surgical personnel.

Treatment success is defined as the absence of any clinical signs of nasolacrimal duct obstruction: presence of epiphora, increased tear film, or mucous discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - < 48 months
* Parent/guardian has the ability to complete a written questionnaire
* For patients with two eyes requiring surgery at enrollment: investigator is planning to perform the same type of surgical procedure on both eyes
* Onset of NLDO symptoms and/or signs prior to 6 months chronological age
* Presence of epiphora, increased tear film, and/or mucopurulent discharge in the absence of an upper respiratory infection or an ocular surface irritation
* Undergoing primary NLDO surgery

Exclusion Criteria:

* History of nasolacrimal duct surgery including simple probing, nasolacrimal intubation, balloon catheter dilation, or dacryocystorhinostomy
* Glaucoma present
* Corneal surface disease

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 973 (Actual)
Dates: Start 2005-02; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael X. Repka, M.D., Study Chair — Wilmer Eye Institute; David I. Silbert, M.D., Study Chair — Family Eye Group
Locations (2):
- United States (2):
  - Wilmer Eye Institute, Baltimore, Maryland
  - Family Eye Clinic, Lancaster, Pennsylvania

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group; Repka MX, Chandler DL, Beck RW, Crouch ER 3rd, Donahue S, Holmes JM, Lee K, Melia M, Quinn GE, Sala NA, Schloff S, Silbert DI, Wallace DK. Primary treatment of nasolacrimal duct obstruction with probing in children younger than 4 years. Ophthalmology. 2008 Mar;115(3):577-584.e3. doi: 10.1016/j.ophtha.2007.07.030. Epub 2007 Nov 8. PMID 17996306
- [Background] Pediatric Eye Disease Investigator Group; Repka MX, Melia BM, Beck RW, Chandler DL, Fishman DR, Goldblum TA, Holmes JM, Perla BD, Quinn GE, Silbert DI, Wallace DK. Primary treatment of nasolacrimal duct obstruction with balloon catheter dilation in children younger than 4 years of age. J AAPOS. 2008 Oct;12(5):451-5. doi: 10.1016/j.jaapos.2008.07.001. PMID 18929305
- [Derived] Miller AM, Chandler DL, Repka MX, Hoover DL, Lee KA, Melia M, Rychwalski PJ, Silbert DI; Pediatric Eye Disease Investigator Group; Beck RW, Crouch ER 3rd, Donahue S, Holmes JM, Quinn GE, Sala NA, Schloff S, Wallace DK, Foster NC, Frick KD, Golden RP, Lambert SR, Tien DR, Weakley DR Jr. Office probing for treatment of nasolacrimal duct obstruction in infants. J AAPOS. 2014 Feb;18(1):26-30. doi: 10.1016/j.jaapos.2013.10.016. PMID 24568978